CLINICAL TRIAL: NCT05140707
Title: The Effect of Virtual Reality on Pain, Anxiety, and Vital Signs of Oncology Patients Undergoing Port Catheter Implantation: A Randomized Controlled Study
Brief Title: Effect of Virtual Reality on Pain, Anxiety, and Vital Signs of the Patients Undergoing Port Catheter Implantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Runida Dogan, Assistant Professor, Inonu University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: VRonPainAnxietyVitalSigns
Record Dates: First submitted 2021-11-08; First posted 2021-12-01 (Actual); Last update posted 2021-12-01 (Actual); Status verified 2021-11

CONDITIONS: Pain; Anxiety; Blood Pressure; Body Temperature Changes
MeSH Terms: conditions — Pain; Anxiety Disorders; Body Temperature Changes

STUDY DESIGN:
Intervention Model Description: The study was of a randomized controlled design. There were two groups in the study; intervention and control. For the intervention group, the virtual reality distraction method was administered to the patients during the port catheter implantation in the intervention group while it wasn't administered to the patients in the control group.
Who Masked: Participant
Masking Description: There wasn't a masking in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): For the patients in this group, a virtual reality device was provided to the patients and patients wear it during the port catheter implantation and after the port catheter implantation when they felt pain.
  Interventions: Other: Virtual Reality Distraction
- Control (No Intervention): For the patients in this group, there wasn't any specific intervention during or after the port catheter implantation.

INTERVENTIONS:
Other: Virtual Reality Distraction — The patients were administered to use the virtual reality device and they were free to choose the theme and video in the library to watch. Patients used the device during the port catheter implantation and untill the 4 hour after the implantation when they felt pain.
  Arms: Intervention

SUMMARY:
This study aimed to determine the effect of virtual reality on pain, anxiety, and vital signs of oncology patients undergoing port catheter implantation. The study was carried out with 139 participants (69 intervention, 70 control) between September 2019 and January 2020. A patient identification form, state anxiety inventory, a table for vital signs, and a visual analog scale for pain severity were used for the data collection. Data were collected from the patients before, during, and after the implantation. In the intervention group, a virtual reality device, movies, and relaxing music were provided to the patients.

DETAILED DESCRIPTION:
To determine the effect of virtual reality (VR) on pain, anxiety, and vital signs of oncology patients undergoing port catheter implantation. The study was a randomized controlled study. The study was carried out with 139 participants (69 intervention, 70 control) between September 2019 and January 2020. Data were collected before, during, and after the implantation by using a patient identification form, State Anxiety Inventory (SAI), a table for vital signs, and a visual analog scale for pain severity. In the intervention group, a virtual reality device, movies, and relaxing music were provided and patients were instructed to use it during the implantation and when they felt pain after the implantation. Data of the study were analyzed with IBM SPSS v25.0.

ELIGIBILITY:
Inclusion Criteria:

* aged 18 years and older, can communicate in Turkish, being diagnosed with cancer, and undergoing port catheter implantation.

Exclusion Criteria:

* being have chronic pain or anxiety disorders, using any type of analgesic or anxiolytic, and diagnosed with epilepsy were excluded from the study. The patients who have a visual impairment or also excluded from the study. Patients diagnosed with brain cancer or have brain metastasis were excluded from the study considering the potential seizures. During the intervention, the interventions were ended for the patients who experienced headache or dizziness (two most common problems caused by VR) and data of these patients were not included in the analysis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
Pain Severity | Change from baseline pain severity at 4 hours
  A visual analog scale was used the examine the pain of the patients. Patients mark the severity of their experiences on 10 cm lines and the beginning of the line shows the lowest degree of the experience while the end of the line shows the highest. This scale is frequently used to determine the severity of the patient's pain. In this study, a 10 cm line was used to assess the severity of the patient's pain. While 0 reflects no pain, 10 reflects the highest severity of the pain. VAS was used for both groups before and after the port catheter implantation.
Anxiety | Change from baseline anxiety levels at 4 hours
  State anxiety inventory was used to examine the patients' anxiety. The scale was by Spielberger et al (1970). The Cronbach's Alpha internal consistency coefficients were range between .83 and .87. The State Anxiety Scale is a 20-item scale about how an individual feels at the moment. Originally, the scale consisted of two main domains, state anxiety, and trait anxiety. Only one of these two domains, state anxiety, was used in this study. The scores on the scale range between 20 and 80. Higher points reflect higher levels of anxiety. The scale was reported valid and reliable for Turkish society. The Cronbach's Alpha of the Turkish version was reported between 0.94 and 0.96. The scale was used for both groups before and after the port catheter implantation.
Blood Pressure (Systolic and Diastolic) | Change from the baseline blood pressure at 4 hours
  The blood pressure of the patients was assessed by using the Con-Tec CMS5100 device. The results presented as mmHg. The blood pressure measuring was administered for the patients in both groups.
Heart Rate | change from baseline heart rate at 4 hours
  Heart rates were assessed by using the Con-Tec CMS5100 device. Beat per minute was used for comparison. Heart rates were measured for both groups.
Respiratory Rate | change from baseline respiratory rate at 4 hours
  The respiratory rate was assessed by using the Con-Tec CMS5100 device. Respiration (inhalation and exhalation) per minute was used for comparison. The respiratory rate was measured for both groups.
O2 saturation | change from baseline O2 saturation at 4 hours
  O2 saturation was assessed by using the Con-Tec CMS5100 device. O2% were used for comparison. O2 Saturation was measured for both groups.

CONTACTS AND LOCATIONS:
Overall Officials: Tuğba Menekli, Ph.D., Study Director — Tuğba Menekli
Locations (1):
- İnönü Üniversitesi, Malatya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No